CLINICAL TRIAL: NCT02645617
Title: Phase 1 Safety Evaluation of Advantage Anti-Caries Varnish
Brief Title: Safety Evaluation of Advantage Anti-Caries Varnish
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advantage Dental Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PVP-I Varnish
Record Dates: First submitted 2015-12-28; First posted 2016-01-05 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Paint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varnish (Experimental): Dental varnish containing povidone iodine and sodium fluoride
  Interventions: Drug: Varnish

INTERVENTIONS:
Drug: Varnish — Topical application to the teeth
  Other Names: Advantage Anti-Caries Varnish

SUMMARY:
The purpose of the study is to confirm the safety of Advantage Anti-Caries Varnish.

DETAILED DESCRIPTION:
This is an open-label Phase 1 study. The active ingredients are Povidone Iodine and Sodium Fluoride [Therametrics Technologies, Inc, Noblesville, IN, USA]. The oral soft tissues and teeth of the children will be examined and the test varnish to the teeth. The child will be re-examined at 24-48 hours for the presence of adverse oral soft tissue changes. At the follow-up, a qualified dental provider will ask questions focused on adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Weight less than 15 kg or hypersensitivity to iodine

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — Advantage Dental
Locations (1):
- University of Washington Regional Clinical Dental Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varnish
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Varnish
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue
Description: Proportion of participants with any oral ulcerations OR inflammatory response
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Varnish
Number analyzed (Participants) | 12
Participants | 0

2. Secondary Outcome: Adverse Events
Description: Proportion of participants with any emergency medical care OR report of nausea OR not eating OR vomiting OR difficulty swallowing OR swelling around the mouth OR itchiness around the mouth OR hives OR rash OR stomach ache OR diarrhea
Time Frame: within 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Varnish
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Intraoral erythema
Arm/Group | Varnish
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No